CLINICAL TRIAL: NCT01091207
Title: A Phase II Study of Sorafenib in Patients With Metastatic or Advanced Gastrointestinal Stromal Tumors Who Failed to Imatinib and Sunitinib
Brief Title: Sorafenib for Imatinib/Sunitinib-failed GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean GIST Study Group (Unknown)
Responsible Party: Se Hoon Park, Samsung Medical Center, Seoul, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-08-102
Record Dates: First submitted 2009-11-30; First posted 2010-03-23 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Sorafenib; GIST; Refractory; advanced GIST failed after both imatinib and sunitinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Experimental): The patients will receive daily oral administration of sorafenib 400 mg twice daily.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — The patients will receive daily oral administration of sorafenib 400 mg twice daily.

SUMMARY:
With discovery of KIT (CD117) mutations and the advent of KIT tyrosine kinase inhibitor imatinib, there has been substantial improvement in overall survival in patients with advanced and/or metastatic gastrointestinal tumors (GIST). Recently, sunitinib showed activity as second-line therapy in GIST patients after failure with imatinib. However, virtually all patients will eventually progress or become intolerable after imatinib and sunitinib. In preclinical models, sorafenib inhibits KIT activity and cell growth of imatinib-resistant tumors. The objective of this multi-center, non-randomized phase II study is to evaluate the safety and activity of sorafenib given as third-line therapy for GIST.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, multi-center, phase II study recruiting patients with advanced GIST who are pretreated with both imatinib and sunitinib. The current study will provide an estimate of the activity and safety of sorafenib in GIST. The primary study endpoint is the disease control rate (DCR), defined as complete or partial response or stable disease of at least 24 weeks of sorafenib therapy. Secondary endpoints include PFS, OS and safety.

Patients with advanced (unresectable and/or metastatic) GIST who failed after previous therapy involving both imatinib and sunitinib will be eligible. Failure to imatinib and sunitinib is defined as disease progression regardless of intervening response during therapy, or intolerance. There is no limit to the number of prior therapies a patient may have received (e.g., patients may have received therapy with nilotinib, other TKIs, or chemotherapy in addition to imatinib or sunitinib).

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* advanced GIST
* failed (progressed and/or intolerable) after prior treatments for GIST
* ECOG performance status of 0~2
* resolution of all toxic effects of prior treatments
* no prior radiotherapy within 1 month before registration
* measurable lesion as defined by RECIST
* adequate marrow, hepatic, renal and cardiac functions
* provision of a signed written informed consent

Exclusion Criteria:

* severe co-morbid illness and/or active infections
* pregnant or lactating women
* history of other malignancies
* active CNS disease not controllable with radiotherapy or corticosteroids
* active and uncontrollable bleeding from gastrointestinal tract
* prior history of sorafenib use
* gastrointestinal obstruction or malabsorption syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Disease-control rate | Six months after registration

SECONDARY OUTCOMES:
Response rate | Every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park SH, Ryu MH, Ryoo BY, Im SA, Kwon HC, Lee SS, Park SR, Kang BY, Kang YK. Sorafenib in patients with metastatic gastrointestinal stromal tumors who failed two or more prior tyrosine kinase inhibitors: a phase II study of Korean gastrointestinal stromal tumors study group. Invest New Drugs. 2012 Dec;30(6):2377-83. doi: 10.1007/s10637-012-9795-9. Epub 2012 Jan 25. PMID 22270258